CLINICAL TRIAL: NCT05203562
Title: The Prophylactic Role of Aromatase Inhibitor Letrozole in Decreasing the Incidence of Gestational Trophoblastic Neoplasia in Patients With Complete Hydatidiform Mole
Brief Title: Letrozole as a Prophylaxis From GTN for Complete Mole Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed Ali Alabiad, MD, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LETROZOLE IN CHM
Record Dates: First submitted 2022-01-19; First posted 2022-01-24 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Gestational Trophoblastic Disease
Keywords: Aromatase Inhibitor; Letrozole; GTN; Complete Mole
MeSH Terms: conditions — Gestational Trophoblastic Disease; Hydatidiform Mole | interventions — Vacuum Curettage; Letrozole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group I (Active Comparator): Patients with complete mole treated by evacuation of using suction curettage followed by conservative follow up
  Interventions: Procedure: Suction evacuation
- Prophylactic letrozole group II (Experimental): Patients with complete mole treated by evacuation of using suction curettage followed by 5mg daily letrozole for 10 days followed by conservative follow up
  Interventions: Procedure: Suction evacuation; Drug: Letrozole tablets

INTERVENTIONS:
Procedure: Suction evacuation — both groups underwent complete mole evacuation using suction curettage.
  Other Names: Evacuation of CHM using Suction curettage
Drug: Letrozole tablets — Group II Patients received 5mg(2tablets 2.5gm) daily letrozole for 10 days after complete mole evacuation
  Other Names: 5mg daily (2 tablets 2.5 gm)
  Arms: Prophylactic letrozole group II

SUMMARY:
Prophylactic use of aromatase inhibitor is effective in decreasing the incidence of Gestational Trophoblastic Neoplasia (GTN) in patients with complete hydatidiform mole (CHM)

DETAILED DESCRIPTION:
Management of hydatidiform mole is usually evacuation followed by β-hcg surveillance to early detect cases of GTN . The risk of developing GTN is reported to be 16% to 20% in women with CHM . GTN is a potentially life-threatening malignancy but has an excellent cure rate. Trials were conducted to assess the role of prophylactic chemotherapy to prevent the development of GTN. In addition to their side effects, a meta-analysis concluded that there is insufficient evidence to support the use of prophylactic chemotherapy in clinical practice. Third-generation aromatase inhibitors such as letrozole have been shown to successfully block estrogen production in women of reproductive age. Their safety, high tolerability, low cost, and associated minimal adverse effects have all been established over several decades of clinical use and recently used successfully alone in the medical treatment of ectopic pregnancy making marked degenerative effects on the placenta.

The study hypothesizes that by inhibiting the estrogen synthetase (the aromatase enzyme) progesterone would not exert its physiological role in maintaining early pregnancy including complete hydatidiform mole. Thus, using a prophylactic aromatase inhibitor after CHM may have a role in the prevention of GTN and more effective clearance of β-hcg.

Rational GTN is a potentially life-threatening malignancy. The risk of progression of CHM to GTN is 20%. Prophylactic use of aromatase inhibitor may decrease the incidence of GTN.

Research question:

Is prophylactic use of aromatase inhibitor effective in decreasing the incidence of GTN in patients with CHM

Hypothesis Prophylactic use of aromatase inhibitor is effective in decreasing the incidence of GTN in patients with CHM

Aim of this work The study aims at figuring out whether prophylactic use of aromatase inhibitor is effective in decreasing the incidence of GTN in patients with CHM.

OBJECTIVES

* To assess the incidence of GTN after the evacuation of CHM without prophylactic use of aromatase inhibitor.
* To assess the incidence of GTN after the evacuation of CHM without prophylactic use of aromatase inhibitor.
* To assess the side effects of aromatase inhibitor when used as a prophylaxis against GTN development in CHM cases.

PATIENTS AND METHODS

Technical design:

* Setting: Department of Obstetrics and Gynecology
* Sample size: 200 patients diagnosed to have CHM by ultrasound and confirmed by histopathological examination.

Operational design:

* Type of the study: a randomized controlled trial.
* Steps of performance and techniques that will be used

women included in the study will be subjected to the following

Preoperative

1. Complete history taking.
2. General and abdominal examination.
3. Routine preoperative laboratory investigations.
4. Ultrasound to diagnose complete hydatidiform mole.
5. Measurement of β-hcg level. Intraoperative

   * Evacuation of CHM using Suction curettage.
   * Tissues obtained during an evacuation will be sent for histological assessment. Post-operative
   * Women will be randomized classified into two groups
   * Control group I: Conservative follow up
   * Prophylactic letrozole group II 5-mg Letrozole will be administered as two 2.5-mg tablets every day for 10 days.
   * All Patients will receive instruction to return for β-hcg follow up which will be done weekly till complete resolution then monthly for 6 months.
   * Participants will be advised to receive contraception during the follow-up period.
   * The patients who will develop GTN in either group will be picked up and the incidence of GTN will be calculated in each group.

ELIGIBILITY:
Inclusion Criteria:

* Women were diagnosed to have CHM by ultrasound and confirmed by histopathological examination

Exclusion Criteria:

* Metastatic disease associated with HM at presentation, in which situation chemotherapy, rather than prophylactic treatment, as prescribed,
* Late diagnosis of CHM made only by histological examination of curetted material
* Uterine evacuation at another hospital and patient seen at the optimum patient care only for follow up

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients with complete hydatidiform mole
Enrollment: 200 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
(β-hCG) level | at the first day of evacuation
  A quantitative human chorionic gonadotropin
(β-hCG) level | one month after evacuation
  A quantitative human chorionic gonadotropin
(β-hCG) level | two months after evacuation
  A quantitative human chorionic gonadotropin
(β-hCG) level | three months after evacuation
  A quantitative human chorionic gonadotropin
(β-hCG) level | four months after evacuation
  A quantitative human chorionic gonadotropin
(β-hCG) level | Five months after evacuation
  A quantitative human chorionic gonadotropin
(β-hCG) level | Six months after evacuation
  A quantitative human chorionic gonadotropin

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Alabiad, MD, Principal Investigator — Zagazig University
Locations (1):
- Mohamed ALI Alabiad, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
3 months after final complete
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months after final complete
Access Criteria: Contac dr Mohamed at drno99@yahoo.com
URL: http://www.staffdata.zu.edu.eg/ar/ShowData/23528